CLINICAL TRIAL: NCT04928183
Title: The Impact of Carbon Monoxide and Altitude on Vascular Function
Acronym: CarMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00096251
Record Dates: First submitted 2021-05-06; First posted 2021-06-16 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2021-06

CONDITIONS: Vasodilation; Vasoconstriction
MeSH Terms: conditions — Aneurysm | interventions — Nitroprusside; Phenylephrine

STUDY DESIGN:
Intervention Model Description: Participants will partake in both room air and CO exposure on 2 separate visits.
Who Masked: Participant
Masking Description: Participant will not be aware of which rebreathe treatment (CO or Room Air) they are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room Air Rebreathe (Sham Comparator): Rebreathe protocol will be completed with a room air syringe rather than CO
  Interventions: Drug: Sodium Nitroprusside; Drug: Phenylephrine Hydrochloride
- CO Rebreathe (Experimental): Rebreathe protocol will be completed with Carbon Monoxide
  Interventions: Other: Carbon monoxide rebreathe; Drug: Sodium Nitroprusside; Drug: Phenylephrine Hydrochloride

INTERVENTIONS:
Other: Carbon monoxide rebreathe — Carbon monoxide exposure to increase blood (Carboxyhemoglobin) COHb safely to ~10%
  Other Names: Schmidt-Prommer blood volume test
  Arms: CO Rebreathe
Drug: Sodium Nitroprusside — Bolus Sodium Nitroprusside (SNP) injection for endothelium-independent vasodilation measure
  Other Names: Nipride
Drug: Phenylephrine Hydrochloride — Bolus Phenylephrine injection for observe α1-mediated vasoconstriction during mild exercise

SUMMARY:
The CarMA (Carbon Monoxide and Altitude) Study aims to observe the vascular effects of carbon monoxide exposure at low and high altitudes.

DETAILED DESCRIPTION:
Each year, millions of people make journeys from low altitude regions to high altitude for recreation, travel, and religious pilgrimage. Carbon monoxide (CO) is commonly associated with cigarette smoke, exhaust fumes, and is viewed as a life-threatening toxic gas. Exposure to CO occurs during travel to and during activities common in high-altitude travel and pilgrimage including vehicle fumes, incense, and second-hand smoke exposure. High altitude exposure and CO exposure have been observed independently to have complex and opposing effects on vascular endothelial function. Observation of these stimuli together in a controlled environment may allow for further understanding of the underlying mechanisms of vascular physiology and adaptations to both high-altitude and CO exposure. The CarMA (Carbon Monoxide and Altitude) Study aims to observe the vascular effects of carbon monoxide exposure at low and high altitudes. Recently, other studies have showed a significant improvement in flow mediated dilation (FMD) with acute exposure to low levels of CO To date, no research has been presented concerning the effect of CO on vascular function at altitude. The present study aims to observe the effect of acute carbon monoxide exposure on 1) flow mediated dilation, 2) conduit artery flow in exercise induced reactive hyperemia at sea level and at altitude, and 3) the effect of CO on vascular function in a high altitude dwelling (sherpa) population.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-50 years
* No medical history of cardiovascular, respiratory, nervous system, or metabolic disease.
* Women must be pre-menopausal.

Exclusion Criteria:

* Participants with any known cardiovascular, respiratory, nervous system, or metabolic disease.
* Having travelled above 2,000m within 1 month of testing at low and high altitude.
* Women who are pregnant, confirmed by a pregnancy test.
* Women who are post-menopausal.
* Participants that are classified as obese (body mass index > 30 kg/m2).
* Participants who are current daily smokers.
* Participants that are currently taking monoamine (MAO) inhibitors, or tricyclic antidepressants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Change in brachial artery diameter (assessed via ultrasound) following release of arterial occlusion | 15 minutes
  Change in brachial artery diameter (assessed via ultrasound) following release of arterial occlusion
Blood flow within the brachial artery during rhythmic handgrip exercise. | 15 minutes
  Blood flow within the brachial artery during rhythmic handgrip exercise.
Change in brachial artery conductance following an infusion of phenylephrine | 5 min
  Change in brachial artery conductance following an infusion of phenylephrine

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, MSc, Principal Investigator — University of Alberta; Craig Steinback, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Basnyat B. High altitude pilgrimage medicine. High Alt Med Biol. 2014 Dec;15(4):434-9. doi: 10.1089/ham.2014.1088. PMID 25330393
- [Background] Rezk-Hanna M, Mosenifar Z, Benowitz NL, Rader F, Rashid M, Davoren K, Moy NB, Doering L, Robbins W, Sarna L, Li N, Chang LC, Elashoff RM, Victor RG. High Carbon Monoxide Levels from Charcoal Combustion Mask Acute Endothelial Dysfunction Induced by Hookah (Waterpipe) Smoking in Young Adults. Circulation. 2019 May 7;139(19):2215-2224. doi: 10.1161/CIRCULATIONAHA.118.037375. PMID 30764644
- [Background] Choi BG, Lee J, Kim SW, Lee MW, Baek MJ, Ryu YG, Choi SY, Byun JK, Mashaly A, Park Y, Jang WY, Kim W, Choi JY, Park EJ, Na JO, Choi CU, Lim HE, Kim EJ, Park CG, Seo HS, Oh DJ, Rha SW. The association of chronic air pollutants with coronary artery spasm, vasospastic angina, and endothelial dysfunction. Coron Artery Dis. 2018 Jun;29(4):336-343. doi: 10.1097/MCA.0000000000000603. PMID 29334505
- [Background] Weber LP, Al-Dissi A, Marit JS, German TN, Terletski SD. Role of carbon monoxide in impaired endothelial function mediated by acute second-hand tobacco, incense, and candle smoke exposures. Environ Toxicol Pharmacol. 2011 May;31(3):453-9. doi: 10.1016/j.etap.2011.02.008. Epub 2011 Feb 26. PMID 21787716
- [Background] Tymko MM, Tremblay JC, Bailey DM, Green DJ, Ainslie PN. The impact of hypoxaemia on vascular function in lowlanders and high altitude indigenous populations. J Physiol. 2019 Dec;597(24):5759-5776. doi: 10.1113/JP277191. Epub 2019 Nov 28. PMID 31677355